CLINICAL TRIAL: NCT05909540
Title: A Prospective Study of Natural History and Clinical Outcomes for Basilar Invagination
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: XW-NS-PNHBI
Record Dates: First submitted 2023-04-02; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-04

CONDITIONS: Basilar Invagination
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Goel A Type Basilar Invagination: 1) ADI>3mm in adults, or ADI>5mm in child.
  Interventions: Procedure: Posterior facet distraction and fusion
- Goel B Type Basilar Invagination: 1. ADI<3mm in adults, or ADI<5mm in child.
  2. The stabilization in atlantoaxial could can be found.
  3. The tip of odontoid can exceed the Chamberlian's line， but not exceed the Wackenheim's line and Mcrae's line.
  Interventions: Procedure: Posterior facet distraction and fusion

INTERVENTIONS:
Procedure: Posterior facet distraction and fusion — With the patient in prone position, cervical traction was only intraoperatively after anesthesia with weights of approximately 5-8 kg during surgery. Monitoring of the spinal cord with motor evoked potential and somatosensory evoked potential were used throughout the surgery. Using a posterior midline incision, the occiput to the C2 spinous process was surgically exposed, separated to the lateral edge of the C1-2 joint, and cut off at the C2 nerve root to expose the C1-2 articular surface Quantitative reduction techniques included the following steps .1) Facet joint release and cage implantation technique 2)Adjusting POCA by cantilever and occipitocervical fixation technique.

SUMMARY:
A Prospective Study of Natural History and Clinical Outcomes for Basilar Invagination

DETAILED DESCRIPTION:
Since basilar invagination was reported, its pathogenesis has been considered both primary and secondary. Surgical treatment methods emerged in an endless stream, and a hundred schools of thought contend. However, the link between the symptoms and imaging has not been studied in detail. We prospectively enrolled patients with basilar depression, and then explored the natural history of the disease and the clinical outcomes of early intervention.

ELIGIBILITY:
Inclusion Criteria:

1. BI discovered by the patient not incidentally;
2. Patients with depression of the skull base caused by congenital skeletal developmental malformations and symptoms;
3. The patient was initially treated in our center, and the interval between onset and treatment was at least 1 month or no treatment;
4. The imaging diagnosis of BI meets the standard (3-5mm higher than the Chamberlain's line)

Exclusion Criteria:

1. secondary BI caused by trauma, pathological factors such as rheumatoid arthritis, hyperparathyroidism, osteogenesis imperfecta, rickets, osteomalacia, spinal cord tumors, tuberculosis, inflammation of adjacent structures, and simple AAD, odontoid body deformity, etc.
2. spinal vascular disease, intervertebral disc herniation, tethered spinal cord disease and other diseases that may cause symptoms.
3. Patients with incomplete imaging data or symptomatic data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with primary basilar depression
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-06 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
improved symptoms | 1 months postoperatively
  The symptoms improved after the opration or natural condition.（JOA scores and SF-12 scores）
improved symptoms | 3 months postoperatively
  The symptoms improved after the opration or natural condition.（JOA scores and SF-12 scores）
improved symptoms | 6 months postoperatively
  The symptoms improved after the opration or natural condition.（JOA scores and SF-12 scores）
improved radiology | 1 months postoperatively
  improved ADI, CCA, CTA ; The basilar invagination reduced
improved radiology | 3 months postoperatively
  improved ADI, CCA, CTA ; The basilar invagination reduced
improved radiology | 6 months postoperatively
  improved ADI, CCA, CTA ; The basilar invagination reduced
operation complication | 1 months postoperatively
  operation complication（Excessive bleeding, bronchopneumonia, vertebral artery injury ）
operation complication | 3 months postoperatively
  operation complication（Excessive bleeding, bronchopneumonia, vertebral artery injury ）
operation complication | 6 months postoperatively
  operation complication（Excessive bleeding, bronchopneumonia, vertebral artery injury ）

CONTACTS AND LOCATIONS:
Overall Officials: Zan Chen, MD. PHD., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital， Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided